CLINICAL TRIAL: NCT02016586
Title: Breastfeeding Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: AL08
Record Dates: First submitted 2013-11-29; First posted 2013-12-20 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-05

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): Subjects in the control group will continue to take the prenatal supplement primarily consisting of folic acid (400 mcg), elemental iron (60 mg) and will receive breastfeeding advice during prenatal visits.
- Intervention (Experimental): Lactation support in conjunction with a maternal nutritional supplement S348S0
  Interventions: Dietary Supplement: Maternal Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: Maternal Nutritional Supplement — S348S0
  Arms: Intervention

SUMMARY:
To evaluate the benefits of a lactation support intervention, in conjunction with maternal nutritional supplementation.

DETAILED DESCRIPTION:
This study aims to evaluate the benefits of a lactation support intervention model combining a maternal nutritional supplementation starting at 8 weeks before delivery to 12 weeks postpartum and a lactation support intervention consisting of 1 prenatal and 3 postnatal sessions on exclusive breastfeeding rate.

ELIGIBILITY:
Inclusion Criteria:

1. Mother with singleton pregnancy at 26 to 29 weeks of gestation.
2. Mother is between 20 and 35 years of age.
3. Mother pre-pregnant BMI < 25.0 kg/m2.
4. Mother is first-time mother.
5. Mother is contactable by telephone.
6. Mother is non-smoker.
7. Infant is a singleton from a full term birth with a gestational age of 37-42 weeks.
8. Infant's birth weight was > 2500 g.
9. Infant is judged to be in good health.
10. Mother confirms her intention to breastfeed and refrain from taking any other nonstudy maternal milk supplement or galactogogues during the study period.

Exclusion Criteria:

1. Mother is allergic or intolerant to any ingredient found in the study product.
2. An adverse maternal, fetal or infant medical history that has potential effects on child's growth and/or development.
3. Mother has gestational diabetes and/or pre-eclampsia.
4. Mother with contraindications to breastfeeding.
5. Gestational weight gain is greater than 14 kg at enrollment.
6. Mother had a breast surgery.
7. Mother and/or newborn infant has major illness that requires intensive care admission.
8. Infant has major congenital anomaly.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2013-11; Primary Completion 2014-10 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Rate | Week 12 postpartum

SECONDARY OUTCOMES:
Breastfeeding Rate | Week 4 postpartum
Lactation Assessment | Week 4 postpartum
  Maternal completed questionnaire with visual analogue scales
Infant Anthropometrics | Week 4 postpartum
  Scale weight; Length and head circumference measurement
Breastfeeding Rate | Week 8 postpartum
Lactation Assessment | Week 8 postpartum
  Maternal completed questionnaire with visual analogue scales
Lactation Assessment | Week 12 postpartum
  Maternal completed questionnaire with visual analogue scales
Infant Anthropometrics | Week 8 postpartum
  Scale weight; Length and head circumference measurement
Infant Anthropometrics | Week 12 postpartum
  Scale weight; Length and head circumference measurement

CONTACTS AND LOCATIONS:
Overall Officials: Dieu Huynh, MD, PhD., Study Chair — Abbott Nutrition
Locations (18):
- Vietnam (18):
  - An Lao District Health Center - Bat Trang, Haiphong
  - An Lao District Health Center - Quoc Tuan, Haiphong
  - An Lao District Health Center - Thai Son, Haiphong
  - An Lao District Health Centre- Quoc Trung, Haiphong
  - An Lao District Health Centre- Truang Tho, Haiphong
  - Bin Luc District Health Centre- Dong Du, Hà Nam
  - Binh Luc District Health Center - An Lao, Hà Nam
  - Binh Luc District Health Center - Binh Nghia, Hà Nam
  - Binh Luc District Health Center - Trang An, Hà Nam
  - Yen Mo District Health Center - Yen Dong, Ninh Bình
  - Yen Mo District Health Center - Yen Hoa, Ninh Bình
  - Yen Mo District Health Center - Yen Thanh, Ninh Bình
  - Phu Binh District Health Center - Kha Son, Thái Nguyên
  - Phu Binh District Health Center - Tan Khanh, Thái Nguyên
  - Phu Binh District Health Center - Tan Kim, Thái Nguyên
  - Phu Binh District Health Centre- Tan Duc, Thái Nguyên
  - Phu Binh District Health Centre- Tan Hoa, Thái Nguyên
  - Phu Binh District Health Centre- Xuan Phuong, Thái Nguyên

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran NT, Nguyen LT, Berde Y, Low YL, Tey SL, Huynh DTT. Maternal nutritional adequacy and gestational weight gain and their associations with birth outcomes among Vietnamese women. BMC Pregnancy Childbirth. 2019 Dec 4;19(1):468. doi: 10.1186/s12884-019-2643-6. PMID 31801514